CLINICAL TRIAL: NCT01954199
Title: The Effectiveness of Neurodynamic Techniques in Patients With Nerve-Related Leg Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Giovanni Esteves Ferreira, Mr, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFCSPA
Record Dates: First submitted 2013-09-24; First posted 2013-10-01 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Nerve Pain; Peripheral Nerve Injuries; Peripheral Nervous System Diseases; Sciatica; Low Back Pain; Low Back Ache; Signs and Symptoms
Keywords: Sciatica; Nerve pain; Low back pain
MeSH Terms: conditions — Neuralgia; Peripheral Nerve Injuries; Peripheral Nervous System Diseases; Sciatica; Low Back Pain; Signs and Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neurodynamic group (Experimental): Patients allocated to this group will receive three different neurodynamic techniques: a lumbar foramen dynamic opener; a side-lying slider and a slider in the slump position. Patients will be asked to perform home exercises (a slider and a tensioner technique). Treatment will receive four treatments during two weeks (two sessions/week).
  Interventions: Procedure: Neurodynamic Group
- Control Group (No Intervention): Patients allocated to Control Group (CG) will receive no intervention and will be advised according to the best evidence available; i.e, advice to remain active and to resume activities of daily living
  Upon trial completion, treatment will be offered.

INTERVENTIONS:
Procedure: Neurodynamic Group — All techniques will be executed in a pain-free way (grade III). Mild discomfort will be accepted, but it must subside as soon as the technique ends.
  * In the dynamic opener technique, patient will be positioned in side-lying, with the affected side upwards. The therapist will then perform grade III oscillations aiming to open the lumbar foramen;
  * In the side-lying slider, the patient will be in side-lying with the affected side upwards. A combination of knee and hip flexion and extension movements will produce sliding in the neural structures;
  * In the slump slider, the patient will be seated in slump position. Combinations between neck and knee movements will produce greater nerve excursion than the side-lying slider. Patients will perform the slump slider in a pain-free manner.
  Other Names: Neural mobilization; Sliders; Tensioners; Nerve tissue management
  Arms: Neurodynamic group

SUMMARY:
This study aims to verify if patients with nerve-related leg pain benefits from neurodynamic treatment over two weeks.

DETAILED DESCRIPTION:
Nerve-related leg pain (NRLP) although less prevalent than low back pain itself, is associated with higher economic and social burden, and has been considered a predictor of chronicity and disability among subjects with low back pain.

Numerous approaches are proposed for its management; however, evidence regarding the best therapeutic approach is lacking. Neurodynamic techniques are proposed to be effective to manage NRLP.

Thus, this study aims to verify, through a randomized controlled trial, the effectiveness of a two-week program of neurodynamic techniques on pain and disability in individuals with NRLP.

ELIGIBILITY:
Inclusion criteria:

* unilateral leg pain (Intensity ≥ 3)
* Pain distal to the buttocks
* Reproduction of symptoms and change in symptoms with structural differentiation (cervical return to neutral position or ankle dorsiflexion) with slump test;

Exclusion criteria:

* cauda equina syndrome;
* bilateral leg pain;
* crossed Lasègue sign;
* previous surgery in the lumbar spine;
* inflammatory arthropathies;
* malignancy
* being in litigation or in work-compensation due to back and/or leg pain
* being receiving physiotherapy treatment at the time of baseline assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Leg Pain Intensity | Two weeks after randomization
  Leg Pain will be measured by a 0-10 Numeric Rating Scale (Pain NRS)
Disability | Two weeks after randomization
  Disability will be measured by the Oswestry Disability Index (ODI)

SECONDARY OUTCOMES:
Leg pain Intensity | Four weeks after randomization
  Leg Pain will me measured by a 0-10 Pain NRS
Disability | Four weeks after randomization
  Disability will be measured by the Oswestry Disability Index (ODI)
Back pain intensity | Two weeks after randomization
  Back Pain will me measured by an 0-10 Pain NRS
Back pain intensity | Four weeks after randomization
  Back Pain will me measured by an 0-10 Pain NRS
Distribution of Symptoms | Two weeks, Four weeks after randomization
  Distribution of symptoms will me measured by a body diagram
Function | Two weeks, Four weeks after randomization
  Function will be measured by the Patient-Specific Functional Scale (PSFS)
Global Perceived Effect | Two weeks, Four weeks after randomization
  Global Perceived Effect will be measured by an 11-point (-5 to +5) Global Perceived Effect Scale

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo F Silva, PhD, Study Chair — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Ferreira G, Stieven F, Araujo F, Wiebusch M, Rosa C, Plentz R, Silva M. Neurodynamic treatment did not improve pain and disability at two weeks in patients with chronic nerve-related leg pain: a randomised trial. J Physiother. 2016 Oct;62(4):197-202. doi: 10.1016/j.jphys.2016.08.007. Epub 2016 Aug 24. PMID 27634158